CLINICAL TRIAL: NCT07121660
Title: Post-operative Changes in Children With Severe Neurological Impairment
Brief Title: Post-operative Changes Study
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other); Canuck Place Children's Hospice Research Initiative (Unknown)
Responsible Party: Principal Investigator, Harold Siden, Dr. Hal Siden, MD, FRCPC, University of British Columbia
Other Study IDs: H24-01880
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Post-operative Functional Decline; Severe Neurological Impairment
Keywords: Severe Neurological Impairment; Post-operative functional decline; Neuroinflammation
MeSH Terms: conditions — Neurologic Manifestations; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will be collecting blood samples from study participants at 6 time points and control participants at 3 time points. A 3 mL aliquot of blood will be collected from participants, via venipuncture at timepoints 1, 3, 4, 5, and 6; and via peripheral line at timepoint 2 and 3 (when venipuncture is not conducted). Additionally, 50uL of blood will be collected from study participants through capillary sampling at timepoint 1.
  Following collection, the samples will be transferred to heparin-coated collection tubes, after which they will be transported to the BC Children's Hospital BioBank for storage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Participants: The study participants are the children with severe neurological impairment (SNI) undergoing major (>90 minute procedure) orthopedic surgery to manage musculoskeletal pathology between the ages of 5 and 18 at the time of surgery and their parent/caregiver. Blood will be collected from the child with SNI (at 6 different time points: at the pre-operative assessment, at the time of surgery, 12-24 hours post-operative, 1-2 weeks post-operative, 6 weeks post-operative and 6 months post-operative). The parent/caregiver of the child will be completing the Caregivers Priorities and Child Health Index of Life with Disabilities (CPCHILD) Questionnaire and answer two supplemental questions (at the pre-operative visit, at a 6-weeks post-operative visit and a 6-month post-operative visit). At the initial pre-operative study visit, the parent/caregiver will also complete a demographics form in which demographic information of the child and the parent/caregiver will be collected.
- Control Participants: The control participants group will consist of neurotypically developing children undergoing spine surgery for scoliosis between the ages of 5 and 18 at the time of their surgical procedure. The child or the parent/caregiver of the child, depending on the age of the child, will complete a demographic form and then have blood samples collected at 3 timepoints (during surgery, 12-24 hours post-operative and 6 months post-operative)

SUMMARY:
The goal of this observational pilot study is to evaluate the feasibility and acceptability of the protocol to explore the functional post-operative trajectory in a developmentally and neurologically impaired pediatric population.

The main objectives of the study are:

* Objective 1: To evaluate the feasibility and acceptability of the study protocol for children and families living with severe neurological impairment (SNI). To evaluate feasibility the investigators will assess consent rate, protocol delivery and outcome completion. To evaluate acceptability, the investigators will conduct end-of-study interviews with caregivers to assess outcomes related to the ease and utility of participating in the study, including the methods of data collection.
* Objective 2: To explore patterns of recovery in children with SNI during the peri-operative period. To do this, the investigators will be be assessing function in children with SNI, quality of life in children with SNI and their families, and the profile of inflammatory biomarkers during the perioperative period. The investigators will then compare the inflammatory profile of these children with SNI against a group of neurotypical children also undergoing surgery. To assess function and quality of life of the child with SNI, the investigators will be using the Caregivers Priorities and Child Health Index of Life with Disabilities (CPCHILD) Questionnaire. Parents/caregivers will also be asked to answer two supplemental questions to provide further insight into 1) other areas of function that were not described by CPCHILD and 2) the quality of life of the caregivers. To collect information on the peri-operative inflammatory profile of the child with SNI and the control participants, the investigators will collect blood samples at different peri-operative time points.

ELIGIBILITY:
Inclusion Criteria for Study Participants

1. Children with severe neurological impairment (SNI), including Gross Motor Function Classification System (GMFCS) levels II, III, IV and V and Communication Function Classification System (CFCS) levels II, III, IV and V, and;
2. undergoing major orthopaedic surgical management of musculoskeletal pathology (spine or hip; major defined as >90 minute procedure with skin-to-skin contact) at the BC Children's Hospital and;
3. between 5 and 18 years at the time of their surgical procedure

Exclusion Criteria for Study Participants:

1. GMFCS level = I and CFCS level = I
2. Non-English-speaking Parents/Caregivers

Inclusion Criteria for Control Group Participants:

1. Neurotypically developing children (GMFCS I and CFCS I) and;
2. undergoing major orthopaedic surgical management of musculoskeletal pathology (spine or hip; major defined as >90 minute procedure with skin-to-skin contact) at the BC Children's Hospital and;
3. Between 5 and 18 years of age at the time of their surgical procedure

Exclusion Criteria for Control Group Participants:

1) Non-English-speaking parents/caregivers

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The BC Children's Hospital Orthopedic Clinic (Hip and Spine) will serve as the main recruitment site.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of the study protocol for children and their families living with severe neurological impairment. | From enrollment to the end-of-study interview approximately 6 months after surgery.
  Feasibility will be assessed using consent rate (the overall average consent rate of children/month), protocol delivery (the percent of on/off protocol children) and outcome completion (the percent of children with complete outcome measures).
To evaluate the acceptability of the study protocol for children and their families living with severe neurological impairment. | From enrollment to the end-of-study interview approximately 6 months after surgery.
  Acceptability will be evaluated using end-of-study interviews with caregivers to assess the ease and utility of participating in the study as it relates to our methods and data collection.

SECONDARY OUTCOMES:
Assess the function in children with SNI, including exploring patterns in specific domains of gain/loss, to explore patterns of recovery in children with severe neurological impairment (SNI) during the peri-operative period. | From enrollment to 6 months following surgery.
  The functional changes of children with SNI over the perioperative period will be assessed using the Caregivers Priorities and Child Health Index of Life with Disabilities (CPCHILD) Questionnaire. The CPCHILD Questionnaire is used to assess the effectiveness of interventions aimed at improving and preserving outcomes for children aged 5-18 years of age with severe disabilities, based on caregivers' perspectives and thus, can be used to track functional changes of children over time. Parents/caregivers will also be asked a supplemental question to provide further insight into other areas of function that were not described by CPCHILD.
Assessing the quality of life in children with SNI and their families, to explore patterns of recovery in children with severe neurological impairment (SNI) during the peri-operative period. | From enrollment to 6 months following surgery.
  This objective will also be assessed using the Caregivers Priorities and Child Health Index of Life with Disabilities (CPCHILD) Questionnaire. The CPCHILD Questionnaire is used to assess the effectiveness of interventions aimed at improving and preserving outcomes for children aged 5-18 years of age with severe disabilities, based on caregivers' perspectives. Within the CPCHILD parents/caregivers are asked questions about their child's quality of life and parents/caregivers will also be asked to answer a supplemental question to provide further insight into the quality of life of caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Siden, Principal Investigator — Department of Pediatrics, UBC; Liisa Holsti, Principal Investigator — Department of Occupational Science and Occupational Therapy, UBC
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
In this small study patient deidentification is a priority and IPD may be a problem for confidentiality.

DOCUMENTS (1):
  • Study Protocol (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT07121660/Prot_000.pdf